CLINICAL TRIAL: NCT05676398
Title: Risk of Cardiac Arrhythmias at Extreme Altitude
Brief Title: Cardiac Arrhythmias at Extreme Altitude
Acronym: SUMMIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2659
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Arrhythmias, Cardiac; Tachycardia, Ventricular; Tachycardia, Supraventricular; Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Tachycardia, Supraventricular; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory rhythm monitoring: Ambulatory rhythm monitoring by use of patch-type device.
  Interventions: Diagnostic Test: Ambulatory rhythm recording

INTERVENTIONS:
Diagnostic Test: Ambulatory rhythm recording — Ambulatory rhythm recording by use of a wearable patch-type device.

SUMMARY:
Background: Exposure to high altitudes has been associated with an increased risk of cardiac arrhythmias in healthy subjects and an increased risk of sudden cardiac death.

Aim: The aim of the present study is to evaluate the risk and the incidence of cardiac arrhythmias at extreme altitude.

Methods: This is a prospective cohort study of healthy volunteers determined to climb Mount Everest. Subjects will be evaluated for eligibility by electrocardiography and echocardiography. All study participants will undergo ambulatory rhythm monitoring in their home environment within 12 weeks of the climb. Subsequently, ambulatory rhythm monitoring will be repeated during the ascent from basecamp to the summit of Mount Everest. The primary endpoint will be the composite of supraventricular and ventricular tachyarrhythmias, and bradyarrhythmias.

DETAILED DESCRIPTION:
Background: Several physiological changes at high altitude give rise to a pro-arrhythmic milieu. A fall in atmospheric pressure at high altitude decreases the partial pressure of oxygen (PaO2) and causes arterial hypoxemia. Respiratory alkalosis secondary to hyperventilation causes hypokalemia and hypocalcemia. Both factors facilitate the occurrence of rhythm disturbances, and may be further exacerbated in an adrenergic state with increased epinephrin levels.

Objectives: The primary objective is to investigate the incidence of supraventricular and ventricular tachyarrhythmias, and the incidence of bradyarrhythmias in climbers during the ascent of Mount Everest. The secondary objective is to investigate clinical, electrocardiographic and echocardiographic predictors of cardiac arrhythmias at extreme altitude.

Methods: This is a prospective cohort study of healthy volunteers climbing Mount Everest. Subjects will be evaluated for eligibility by electrocardiography and echocardiography. All participants will undergo a stress test in order to rule out pre-existing rhythm disturbances during exercise. Study participants will undergo ambulatory rhythm monitoring in their home environment within 12 weeks of the climb. Subsequently, subjects will repeat ambulatory rhythm monitoring during the ascent from basecamp to the summit of Mount Everest. The subjects will act as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Normal electrocardiogram
* Normal echocardiography
* Written informed consent

Exclusion Criteria:

* Known cardiac arrhythmia
* Evidence of AV-block, left bundle branch block, or repolarization disorders on electrocardiogram
* Evidence of structural heart disease (valve disease more than mild) or compromised left ventricular ejection fraction as assessed by echocardiography
* Symptoms or history of skin cancer, rash, skin disease, keloid or injury
* Cardiac pacemakers, cardiac defibrillators, implantable electrical devices
* Pregnancy, breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers climbing Mount Everest.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants detected to have cardiac arrhythmia | The primary endpoint will be assessed during the ascent from basecamp to the summit of Mount Everest and back to basecamp, expected to be on average 5-10 days.
  Composite of supraventricular and ventricular tachyarrhythmias, and bradyarrhythmias.

SECONDARY OUTCOMES:
Patterns in the occurrence of cardiac arrhythmias | The outcome will be assessed during the ascent from basecamp to the summit of Mount Everest and back to basecamp, expected to be on average 5-10 days.
  Occurrence of the composite of supraventricular and ventricular tachyarrhythmias, and bradyarrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, Principal Investigator — Bern University Hospital, University of Bern, Switzerland
Locations (1):
- National Academy of Medical Sciences, Bir Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No